CLINICAL TRIAL: NCT06012903
Title: Epidemiological Study of Lower Urinary Tract Symptoms and School Functioning in Children in Regular Elementary School
Brief Title: Lower Urinary Tract Symptoms and School Functioning in Children
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Ghent (Other)
Collaborators: University Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: BC-11326
Record Dates: First submitted 2023-07-31; First posted 2023-08-28 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: Lower Urinary Tract Symptoms; Neurodevelopmental Disorders; Incontinence, Urinary; ADHD; ASD; Developmental Coordination Disorder; Child Development; Quality of Life
Keywords: lower urinary tract symptoms; Quality of life; Pediatrics; neurodevelopmental disorders; VSSDES; DCD-Q
MeSH Terms: conditions — Lower Urinary Tract Symptoms; Neurodevelopmental Disorders; Urinary Incontinence; Attention Deficit Disorder with Hyperactivity; Motor Skills Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Parents
  Interventions: Other: Questionnaire Vancouver symptom score for dysfunctional elimination syndrome; Other: Developmental Coordination Disorder Questionnaire; Other: Questionnaire concerning LUTS, NDDs and treatment perceptions
- Children
  Interventions: Other: Questionnaire Welbevinden
- Teachers
  Interventions: Other: Questionnaire about policies and practices regarding children's toilet use and drinking habits in the classroom

INTERVENTIONS:
Other: Questionnaire Welbevinden — A validated questionnaire recommended by the Flemish inspection of education to measure well-being in primary school children of the 4th, 5th and 6th grade.
  Groups: Children
Other: Questionnaire Vancouver symptom score for dysfunctional elimination syndrome — Vancouver symptom score for dysfunctional elimination syndrome, Dutch version, validated by 't Hoen et al. 2016.
  Other Names: VSSDES
  Groups: Parents
Other: Developmental Coordination Disorder Questionnaire — Validated Developmental Coordination Disorder Questionnaire, Dutch version includes assessment of motor functioning.
  Other Names: DCD-Q
  Groups: Parents
Other: Questionnaire concerning LUTS, NDDs and treatment perceptions — Unvalidated, complementary questions including the presence of LUTS, earlier diagnosis of bladder and/or boweldysfunction and neurodevelopmental disorders and perception concerning treatment characteristics.
  Groups: Parents
Other: Questionnaire about policies and practices regarding children's toilet use and drinking habits in the classroom — These unvalidated questionnaire was based on the questionnaire developed by Ko et al. (2016) about the school's policies and practices regarding children's toilet use and drinking habits in the classroom, covering students in grades one through six. Epidemiological questions related to LUTS were added to complement the questionnaire.
  Groups: Teachers

SUMMARY:
Children in primary school often suffer from lower urinary tract symptoms (LUTS), which may negatively impact their overall well-being. Co-occurring neurodevelopmental disorders (NDDs) can adversely affect children as well and can cause restrictions in their daily life, especially in their school-environment.

The goal of this observational study is to identify the prevalence of LUTS in Flemish primary school children.The main questions it aims to answer are:

* How prevalent are LUTS in regular primary education?
* Is there a relation with well-being in school environment?
* Is there an influence of co-occuring NDDs? Children, parents and teachers will be asked to fill in questionnaires related to this research question.

ELIGIBILITY:
Inclusion Criteria:

* Children in 4th-6th grade
* Parents whose children are in grades 1-6
* Teachers responsible for teaching children in grades 1-6
* Children who attend regular primary education
* Capable of speaking & comprehending Dutch

Exclusion Criteria:

* High school students
* home-schooled children
* children who attend special needs education
* Language barrier to understanding Dutch

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children following education in recruited primary, regular education schools and their respective parents/guardians and teachers
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2022-10-06 (Actual); Primary Completion 2025-06-06 (Estimated); Study Completion 2025-06-06 (Estimated)

PRIMARY OUTCOMES:
Bladder and bowel dysfunction | through study completion from the parent-group, 25 minutes
  Prevalence of lower urinary tract symptoms and/or bowel symptoms measured with the vancouver symptom score for dysfunctional elimination syndrome.
School functioning | through study completion from the children-group, 30 minutes
  Quality of life in school environment, measured as the child's well-being about school functioning with the questionnaire Welbevinden.

SECONDARY OUTCOMES:
Influencing factors on school functioning | through study completion from the parent-, children- and teacher-group, 30 minutes
  Prevalence and influence of neurodevelopmental disorders, school-related factors and LUTS. Results from the vancouver symptom score for dysfunctional elimination syndrome, Developmental Coordination Disorder Questionnaire, questions concerning neurodevelopmental disorders and a questionnaire about policies and practices regarding children's toilet use and drinking habits in the classroom will be correlated with results from the questionnaire Welbevinden.
Perception of treatment characteristics | through study completion of the parent-group, 25 minutes
  Perception of parents about treatment characteristics for lower urinary tract symptoms are evaluated by means of a questionnaire including questions about treatment perceptions .

CONTACTS AND LOCATIONS:
Overall Officials: Ellen Vandamme, MD, Principal Investigator — University Hospital, Ghent; Bieke Samijn, PhD, Principal Investigator — University Ghent
Locations (1):
- Ghent University Hospital/Ghent University, Ghent, East Flanders, Belgium

IPD SHARING:
Plan to Share IPD: No